CLINICAL TRIAL: NCT01952340
Title: A Phase II/III, Randomized, Double-Blinded, Controlled Clinical Trial to Investigate the Efficacy of Dietary Flaxseed for the Reduction of Blood Pressure in Newly Diagnosed Hypertensive Individuals
Brief Title: The Efficacy of Dietary Flaxseed for the Reduction of Blood Pressure in Newly Diagnosed Hypertensive Individuals
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Premature termination because: a) the COVID-19 pandemic stopped recruitment or participation for 2 years which limited study numbers, and, b) both PI's will retire and, therefore, will be unable to oversee the trial.
Sponsor: St. Boniface Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Grant Pierce, Executive Director of Research and Professor, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HF2013; B2013:079 (Other: University of Manitoba Research Ethics Board)
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flaxseed (Experimental): 30 grams of milled flaxseed on its own or baked into food products (ie: bagels, muffins, and snack bars)
  Interventions: Dietary Supplement: Flaxseed
- Wheat/Mixed Dietary Oils (Placebo Comparator): A combination of wheat, pecans, and/or mixed dietary oils on its own or baked into food products (ie: bagels, muffins, and snack bars)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Flaxseed — Milled flaxseed
  Arms: Flaxseed
Dietary Supplement: Placebo — Wheat germ/wheat bran and mixed dietary oils
  Arms: Wheat/Mixed Dietary Oils

SUMMARY:
The World Health Organization has deemed high blood pressure as a global crisis because it is the number one risk factor associated with most deaths worldwide. Therefore, the need for effective and desirable treatment options is vitally necessary. The purpose of the current investigation is to determine the efficacy of a new therapeutic strategy: flaxseed. The aim is to determine the efficacy of consuming milled flaxseed every day for 6 months on the reduction of blood pressure in individuals newly diagnosed with high blood pressure yet to receive any blood pressure lowering medications. Secondary objectives are to understand how flaxseed at the molecular level can reduce blood pressure. The study hypothesis is that the flaxseed group will exhibit significant reductions in blood pressure and therefore not require any blood pressure lowering medication. The aim is to provide knowledge on a new therapeutic strategy to help manage high blood pressure.

DETAILED DESCRIPTION:
This trial is a phase II/III, randomized, double-blinded, controlled clinical trial to determine the efficacy of dietary flaxseed as a therapeutic strategy to reduce blood pressure in newly diagnosed hypertensive individuals. The aim of the trial is to recruit 100 participants that have been clinically diagnosed with hypertension within 6 months and yet to receive any anti-hypertensive medication. The control and flax groups will be provided food products to consume on a daily basis for 6 months. Assessment parameters such as averaged automated blood pressure, anthropometrics, 24-food recall, physical activity questionnaire, and blood and urine analysis will be conducted at baseline, 2, 4, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension (average automated systolic blood pressure of 135-160 OR diastolic blood pressure of 85-100)
2. Newly diagnosed. Defined as being clinically diagnosed within the last 6 months. This includes the screening examination.
3. Either gender
4. Untreated for hypertension
5. 18-85 years old and able to provide informed consent.
6. Females who are:

   1. highly unlikely to conceive due to surgical sterilization
   2. postmenopausal female with >2 years since last menses
   3. or non-sterilized, premenopausal female who agrees to: 1. Use an adequate method of contraception to prevent pregnancy (such as a double-barrier method or hormonal); 2. Abstain from heterosexual activity for study period; or 3. Only engage in heterosexual activity with surgically sterilized male partner(s) and not planning on becoming pregnant during the study. Please note that a pregnancy test will NOT be administered for the trial.
7. Subjects taking anti-platelet therapy must be on a stable dose for 3 months prior to the study.
8. Subjects taking lipid lowering drugs must be on a stable dose for 3 months prior to the study.
9. Subjects must have access to freezer space in their residence to hold up to one month of frozen food products associated with this study.

Exclusion Criteria:

1. Patients with ischemic pain at rest in limbs, ulceration, or gangrene.
2. Clinical evidence of peripheral artery disease, previous myocardial infarction, or stroke.
3. Patient has undergone percutaneous coronary angioplasty, has had coronary bypass within the last 6 months, or has unstable angina.
4. Known secondary hypertension of any etiology.
5. Patients with confirmed and clinically significant renal or hepatic abnormalities (creatinine > 0.130 mM or creatinine clearance < 45ml/min, AST 2-3x normal, ALT > 2-3x normal) and/or electrolyte imbalance serum K+ < 3.5 or > 5.5 mM.
6. History of major bleeding.
7. Patients with diabetes mellitus, bowel disease (including Crohn's disease, celiac disease, colitis, peptic ulcer disease, irritable bowel syndrome and diverticulosis) or other diseases such as active systemic lupus erythematosus, cancer, or end stage respiratory disease.
8. Patients with macrovascular target organ damage, including: cerebrovascular disease, stroke, dementia, hypertensive retinopathy, left ventricular dysfunction, angina pectoris, myocardial infarction, renal disease, and peripheral artery disease.
9. Patients with clinical evidence of heart failure or an estimated life expectancy less than 2 years and with high baseline cardiac risk (post ischemic or diabetic cardiomyopathy with an ejection fraction < 40%, Canadian Cardiovascular Society Class 3 or 4 angina or need for coronary revascularization procedures).
10. Subjects that are on supplements other that those prescribed by their clinician for the entire duration of the study. Please see point 11 below.
11. Subjects ingesting more than 2 servings of fish per week, taking omega-3 fatty acid supplements, and/or consuming milled flaxseed or flax oil on a regular basis (ie: ≥ 1 tablespoon of milled flaxseed or 1 teaspoon of flax oil per week). If the patient chooses to, they may exclude these supplements for 4 weeks as a washout period before entry into the trial.
12. Patients having participated in an investigational drug program in the preceding 30 days or unable or unwilling to comply with the protocol.
13. Subjects with allergies to any ingredient in the study product or placebo (including gluten).
14. Patients who will undergo surgery or intend to move well outside Winnipeg during the trial period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
averaged automated blood pressure | Baseline, 2, 4, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Grant N Pierce, Ph.D., Principal Investigator — St. Boniface Hospital Research Centre
Locations (3):
- Canada (3):
  - St. Boniface Hospital Research Centre, Winnipeg, Manitoba
  - South Sherbrook Health Centre, Winnipeg, Manitoba
  - Health Sciences Centre Hospital, Winnipeg, Manitoba

REFERENCES:
- [Background] Rodriguez-Leyva D, Weighell W, Edel AL, LaVallee R, Dibrov E, Pinneker R, Maddaford TG, Ramjiawan B, Aliani M, Guzman R, Pierce GN. Potent antihypertensive action of dietary flaxseed in hypertensive patients. Hypertension. 2013 Dec;62(6):1081-9. doi: 10.1161/HYPERTENSIONAHA.113.02094. Epub 2013 Oct 14. PMID 24126178
- [Derived] Caligiuri SP, Penner B, Pierce GN. The HYPERFlax trial for determining the anti-HYPERtensive effects of dietary flaxseed in newly diagnosed stage 1 hypertensive patients: study protocol for a randomized, double-blinded, controlled clinical trial. Trials. 2014 Jun 18;15:232. doi: 10.1186/1745-6215-15-232. PMID 24938224